CLINICAL TRIAL: NCT05455177
Title: Within-person Change in Patient-reported Outcomes and Their Association With the Wish to Undergo Joint Surgery During a Digital First-line Intervention for Osteoarthritis
Brief Title: Change in Patient Reported Outcomes and Wish for Joint Surgery
Status: Completed | Type: Observational
Sponsor: Joint Academy (Industry)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Other Study IDs: JAPROMS_w
Record Dates: First submitted 2022-06-30; First posted 2022-07-13 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Osteoarthritis, Knee and Hip
Keywords: osteoarthritis; exercise; wish for surgery; digital intervention; PROMs
MeSH Terms: conditions — Osteoarthritis; Motor Activity | interventions — Educational Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Digital first-line intervention for osteoarthritis including exercise and education — The digital OA management programme was delivered by a smartphone application, including education and exercises based on a face-to-face osteoarthritis self-management programme provided nationwide in Sweden and designed according to national and international guidelines. Over 12 weeks, which is the recommended minimum duration of a self-management intervention for OA, a total of 163 exercise sessions and 31 educational sessions are provided.

SUMMARY:
Aim To investigate associations between within-person change in patient reported outcomes (PROMs) and wish for joint surgery during up to 12-month participation in a digital first-line intervention for knee and hip osteoarthritis (OA) comprising exercise and education.

Methods Retrospective observational registry data. All participants enrolling between June 1st 2018 and September 30th 2021 with follow-up data and with a change in their wish for surgery (dichotomous, becoming wishing or unwishing) were included. Analysed PROMS comprised pain (numeric rating scale (NRS), 0-10), 5 level EuroQol - 5-dimension (EQ5D-5L, 0.243-0.976), overall health (NRS, 0-10), activity impairment (NRS, 0-10), walking difficulties (yes/no), fear of movement (yes/no), function and quality of life subscales of Knee/Hip injury and Osteoarthritis Outcome Score 12 Items (KOOS-12/HOOS-12, both 0-100). To capture effects of changes in PROMs over time on probability of wish for surgery, the investigators used fixed effect (conditional) logistic regressions.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of knee or hip osteoarthritis
* Date of enrolment between June 1st 2018 and September 30th 2021 (study period)
* Consent to the use of the data at the moment of enrolment (not withdrawn during the study period)

Exclusion Criteria:

* No follow-up data
* No change in wish for surgery (participants remained either wishing or not wishing to undergo surgery for the whole treatment period). This exclusion was due to the focus of the present study on within-person relationships between PROMs and wish for surgery. In this scenario, those with no change in their wish for surgery do not provide any information to the analysis.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: People with osteoarthritis of the knee or hip ascertained by a clinicians who enrolled in a first-line digital intervention for OA including exercise and education.
Sampling Method: Non-Probability Sample
Enrollment: 14018 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Wish for surgery at baseline | 0 months
  Wish for surgery was monitored by asking the participants 'Are your symptoms so severe that you wish to undergo surgery in your [knee/hip]?' (dichotomous reply, yes/no).
Wish for surgery at 3 months | 3 months
  Wish for surgery was monitored by asking the participants 'Are your symptoms so severe that you wish to undergo surgery in your [knee/hip]?' (dichotomous reply, yes/no).
Wish for surgery at 6 months | 6 months
  Wish for surgery was monitored by asking the participants 'Are your symptoms so severe that you wish to undergo surgery in your [knee/hip]?' (dichotomous reply, yes/no).
Wish for surgery at 9 months | 9 months
  Wish for surgery was monitored by asking the participants 'Are your symptoms so severe that you wish to undergo surgery in your [knee/hip]?' (dichotomous reply, yes/no).
Wish for surgery at 12 months | 12 months
  Wish for surgery was monitored by asking the participants 'Are your symptoms so severe that you wish to undergo surgery in your [knee/hip]?' (dichotomous reply, yes/no).

CONTACTS AND LOCATIONS:
Locations (1):
- Joint Academy, Malmo, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No